CLINICAL TRIAL: NCT04645199
Title: National Longitudinal Cohort of Hematological Diseases (NICHE)
Brief Title: National Longitudinal Cohort of Hematological Diseases
Acronym: NICHE
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: NICHE-cohort
Record Dates: First submitted 2020-11-13; First posted 2020-11-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma; Acute Myeloid Leukemia; Hemophilia; Hemophilia A; Hemophilia B; Myelodysplastic Syndrome; MDS; Lymphoma; Leukemia; Aplastic Anemia; Bleeding Disorder; Bone Marrow Transplantation; Blood Disease Infection; Autoimmune Hemolytic Anemia, AIHA; Essential Thrombocythemia, ET; Large Granular Lymphocyte Leukemia, LGLL; Paroxysmal Nocturnal Hemoglobinuria, PNH
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Myeloid, Acute; Hemophilia A; Hemophilia B; Myelodysplastic Syndromes; Lymphoma; Leukemia; Anemia, Aplastic; Hemostatic Disorders; Anemia, Hemolytic, Autoimmune; Thrombocythemia, Essential; Leukemia, Large Granular Lymphocytic; Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Hematological diseases are disorders of the blood and hematopoietic organs. The current hematological cohorts are mostly based on single-center or multi-center cases, or cohorts with limited sample size in China. There is a lack of comprehensive and large-scale prospective cohort studies in hematology. The purpose of this study is to analyze the incidence and risk factors of major blood diseases, the treatment methods, prognosis and medical expenses of these patients in China.

Method The study will include patients diagnosed with acute myeloid leukemia, multiple myeloma, hemophilia, aplastic anemia, leukemia, myelodysplastic syndrome, lymphoma, bleeding disorders, autoimmune hemolytic anemia, large granular lymphocyte leukemia, essential thrombocythemia, blood infection or received bone marrow transplantation in the investigating hospitals from January 1, 2020, and collect basic information, diagnostic and treatment information, prognosis information, as well as medical expense information from medical records. In its current form, the NICHE registry incorporates historical data (collected from 2000) and is systematically collecting prospective data in two phases with broadening reach, and prospectively follow-up to collect the prognosis information.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with acute myeloid leukemia, multiple myeloma, hemophilia, aplastic anemia, leukemia, myelodysplastic syndrome, lymphoma, bleeding disorders or received bone marrow transplantation in the investigating hospitals from January 1, 2020.

Exclusion Criteria:

* Long-term follow-up information for patients is not available for any reason, such as not being available or having a serious concomitant disease.
* Alcohol and drug addictions affect their ability to comply with study requirements.
* According to the investigator, there are conditions that may endanger the patient's safety or affect his/her compliance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were diagnosed with acute myeloid leukemia, multiple myeloma, hemophilia, aplastic anemia, leukemia, myelodysplastic syndrome, lymphoma, bleeding disorders or received bone marrow transplantation in the investigating hospitals from January 1, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and distribution | 5 years
  To describe the incidence and population characteristics of hematological diseases in China, such as: leukemia, multiple myeloma, hemophilia, aplastic anemia, myelodysplastic syndrome, lymphoma, bleeding disorders, blood disease infection, et al., and analyze the risk factors associated with these diseases.

SECONDARY OUTCOMES:
Therapeutic evaluation | 5 years
  To analyze the therapeutic efficacy and long-term prognosis of patients with hematological diseases, such as: leukemia, multiple myeloma, hemophilia, aplastic anemia, myelodysplastic syndrome, lymphoma, bleeding disorders, blood disease infection, et al.
Health economic evaluation | 5 years
  To conduct health economic evaluation on patients with hematological diseases, such as: leukemia, multiple myeloma, hemophilia, aplastic anemia, myelodysplastic syndrome, lymphoma, bleeding disorders, blood disease infection, et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Lu N, Liu L, Cao Y, Zhang R, Zhai W, Chen X, Ma Q, Yang D, Pang A, Wei J, He Y, Feng S, Han M, Jiang E. Efficacy and safety of mitoxantrone hydrochloride liposome-containing regimens in treating refractory/relapsed acute myeloid leukemia. Discov Oncol. 2025 May 12;16(1):727. doi: 10.1007/s12672-025-02526-y. PMID 40353947
- [Derived] Gao H, Wang J, Zheng X, Pei X, Zheng Y, Zhai W, Zhang R, Chen X, Ma Q, Wei J, Yang D, Pang A, He Y, Feng S, Cao Y, Jiang E. Ursodeoxycholic acid does not reduce SARS-CoV-2 infection in newly allogeneic hematopoietic stem cell transplantation recipients: a prospective NICHE cohort. Front Cell Infect Microbiol. 2024 Mar 5;14:1324019. doi: 10.3389/fcimb.2024.1324019. eCollection 2024. PMID 38505288
- [Derived] Cui J, Yu T, Lv R, Liu J, Fan H, Yan W, Xu J, Du C, Deng S, Sui W, Ho M, Xu Y, Anderson KC, Dong X, Qiu L, An G. Longitudinal genetically detectable minimal residual disease by fluorescence in situ hybridization confers a poor prognosis in myeloma. Ther Adv Med Oncol. 2024 Jan 19;16:17588359231221340. doi: 10.1177/17588359231221340. eCollection 2024. PMID 38249329
- [Derived] Fan H, Wang B, Shi L, Pan N, Yan W, Xu J, Gong L, Li L, Liu Y, Du C, Cui J, Zhu G, Deng S, Sui W, Xu Y, Yi S, Hao M, Zou D, Chen X, Qiu L, An G. Monitoring Minimal Residual Disease in Patients with Multiple Myeloma by Targeted Tracking Serum M-Protein Using Mass Spectrometry (EasyM). Clin Cancer Res. 2024 Mar 15;30(6):1131-1142. doi: 10.1158/1078-0432.CCR-23-2767. PMID 38170583
- [Derived] Yan W, Xu J, Fan H, Li L, Cui J, Du C, Deng S, Sui W, Xu Y, Hao M, Anderson KC, Zou D, Qiu L, An G. Early relapse within 18 months is a powerful dynamic predictor for prognosis and could revise static risk distribution in multiple myeloma. Cancer. 2024 Feb 1;130(3):421-432. doi: 10.1002/cncr.35056. Epub 2023 Oct 17. PMID 37846845
- [Derived] Liu J, Yan W, Fan H, Xu J, Li L, Du C, Mao X, Yan Y, Xu Y, Sui W, Deng S, Yi S, Anderson KC, Qiu L, Zou D, An G. Clinical Benefit of Autologous Stem Cell Transplantation for Patients with Multiple Myeloma Achieving Undetectable Minimal Residual Disease after Induction Treatment. Cancer Res Commun. 2023 Sep 6;3(9):1770-1780. doi: 10.1158/2767-9764.CRC-23-0185. eCollection 2023 Sep. PMID 37680953
- [Derived] Cui J, Lv R, Yu T, Yan W, Xu J, Fan H, Li L, Liu Y, Du C, Deng S, Sui W, Xu Y, Yi S, Zou D, Qiu L, An G. Minor clone of del(17p) provides a reservoir for relapse in multiple myeloma. Haematologica. 2024 Feb 1;109(2):591-603. doi: 10.3324/haematol.2023.283533. PMID 37534514
- [Derived] Fan H, Wang W, Zhang Y, Wang J, Cheng T, Qiu L, Wang X, Xia Z, An G. Current treatment paradigm and survival outcomes among patients with newly diagnosed multiple myeloma in China: a retrospective multicenter study. Cancer Biol Med. 2023 Jan 12;20(1):77-87. doi: 10.20892/j.issn.2095-3941.2022.0612. PMID 36647781

DOCUMENTS (8):
  • Study Protocol: NICHE-AML (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT04645199/Prot_000.pdf
  • Study Protocol: NICHE-MM (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT04645199/Prot_001.pdf
  • Study Protocol: NICHE-Hemophilia (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT04645199/Prot_002.pdf
  • Study Protocol: NICHE-AA (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT04645199/Prot_003.pdf
  • Study Protocol and Statistical Analysis Plan: NICHE-Leukemia/MDS/Lymphoma/BD (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT04645199/Prot_SAP_004.pdf
  • Study Protocol and Statistical Analysis Plan: NICHE-BMT/Pediatrics (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT04645199/Prot_SAP_005.pdf
  • Study Protocol and Statistical Analysis Plan: NICHE-BDI (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT04645199/Prot_SAP_007.pdf
  • Statistical Analysis Plan: NICHE-AA/Hemophilia/AML/MM_SAP (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT04645199/SAP_006.pdf